CLINICAL TRIAL: NCT03760913
Title: OLP-1002 - A First-in-human, Double-blind, Placebo-controlled, Single and Multiple Subcutaneous Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Healthy Male and Female Subjects
Brief Title: OLP-1002 is Being Studied in the Treatment of Pain.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: OliPass Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OLP-1002-001
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: Pain; Pain Injection
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This will be a double-blind, randomized, placebo-controlled, single and multiple subcutaneous dose study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OLP-1002: Part A, Single Ascending Dose (Experimental): Subcutaneous Injection: 30 ng, 120 ng, 400 ng, 1.2 μg, 3 μg, 6 μg, 12 μg, 20 μg, 40 μg, 80 μg, 160 μg
  Interventions: Drug: OLP-1002 (Test): Part A, Single Ascending Dose
- OLP-1002: Part B, Multiple Ascending Dose (Experimental): Subcutaneous Injection: 5 x 2 μg, 5 x 5 μg, 5 x 10 μg, 5 x 20 μg, 5 x 40 μg, 5 x 80 μg
  Interventions: Drug: OLP-1002 (Test): Part B, Multiple Ascending Dose
- Placebo Part A, Single Ascending Dose (Placebo Comparator): Subcutaneous Injection: Placebo
  Interventions: Other: Placebo: Placebo Part A, Single Ascending Dose
- Placebo Part B, Multiple Ascending Dose (Placebo Comparator): Subcutaneous Injection: Placebo x 5
  Interventions: Other: Placebo: Placebo Part B, Multiple Ascending Dose

INTERVENTIONS:
Drug: OLP-1002 (Test): Part A, Single Ascending Dose — Subcutaneous Injection: 30 ng, 120 ng, 400 ng, 1.2 µg, 3 µg, 6 µg, 12 µg, 20 µg, 40 μg, 80 μg, 160 μg
  Arms: OLP-1002: Part A, Single Ascending Dose
Drug: OLP-1002 (Test): Part B, Multiple Ascending Dose — Subcutaneous Injection: 5 x 2 μg, 5 x 5 μg, 5 x 10 μg, 5 x 20 μg, 5 x 40 μg, 5 x 80 μg
  Arms: OLP-1002: Part B, Multiple Ascending Dose
Other: Placebo: Placebo Part A, Single Ascending Dose — Subcutaneous Injection: Placebo
  Arms: Placebo Part A, Single Ascending Dose
Other: Placebo: Placebo Part B, Multiple Ascending Dose — Subcutaneous Injection: Placebo x 5
  Arms: Placebo Part B, Multiple Ascending Dose

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of single and multiple subcutaneous doses of OLP-1002 in healthy subjects.

DETAILED DESCRIPTION:
The exploratory objectives of the study are to evaluate the pharmacodynamic effect of OLP-1002 following single subcutaneous doses in healthy volunteers using a capsaicin pain model, and to monitor the effects of a single subcutaneous doses of OLP-1002 on cardiac QT interval. Where possible, single and/or multiple subcutaneous dose pharmacokinetics of OLP-1002 in healthy subjects will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females of any race, between 18 and 60 years of age, inclusive.
* Body mass index between 18.0 and 28.0 kg/m², inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, single 12-lead electrocardiogram (resting heart rate > 45 bpm and < 90 bpm), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening as assessed by the Investigator (or designee).
* Willing to abide by the contraception requirements.
* Able to comprehend and willing to sign an Informed Consent Form and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* Any of the following:

  * QT interval corrected for heart rate using Fridericia's method > 450 ms confirmed by repeat measurement.
  * QRS duration > 110 ms confirmed by repeat measurement.
  * PR interval > 220 ms confirmed by repeat measurement.
  * findings which would make QT interval corrected for heart rate measurements difficult or QT interval corrected for heart rate data uninterpretable.
  * history of additional risk factors for torsades de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome).
* Female subjects who are pregnant or breastfeeding.
* History of alcoholism or drug/chemical abuse within 1 year prior to Screening.
* Alcohol consumption of > 21 units per week for males and >14 units per week for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
* Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Check-in.
* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* Active skin conditions such as dermatitis, allergy, eczema, psoriasis, or abnormal healing.
* Tattoos, scars, or moles that in the opinion of the Investigator are likely to interfere with dosing or study assessments at any of the potential injection sites.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days or 5 half-lives of the investigational product, whichever is longer, prior to Check-in.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptive concomitant medications within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee) and/or Sponsor have given their prior consent.
* Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
* Receipt of blood products within 60 days prior to Check-in.
* Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
* Poor peripheral venous access.
* Have previously completed or withdrawn from this study or any other study investigating OLP-1002, and have previously received the investigational product.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.
* Part A - PD assessment groups only

  * Subjects considered non-acceptable responders to the intradermal capsaicin test at screening, defined as maximum VAS score of < 3.0 or > 9.0.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Firas Almazedi, MBChB, MSc, CPI, DipPharmMed, Principal Investigator — Covance CRU Leeds
Locations (1):
- Leeds CRU, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Part A, Single Ascending Dose: Placebo: Part A, Single Ascending Dose: Subcutaneous Injection: Placebo
- 30 ng OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 30 ng
- 120 ng OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 120 ng
- 400 ng OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 400 ng
- 1.2 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 1.2 µg
- 3 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 3 µg
- 6 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 6 µg
- 12 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 12 µg
- 20 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 20 µg
- 40 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 40 µg
- 80 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 80 µg
- 160 µg OLP-1002: Part A, Single Ascending Dose: OLP-1002 (Test): Part A, Single Ascending Dose: Subcutaneous Injection: 160 µg
- 5 x Placebo Part B, Multiple Ascending Dose: Placebo: Part B, Multiple Ascending Dose: Subcutaneous Injection: Placebo x 5
- 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose: OLP-1002 (Test): Part B, Multiple Ascending Dose: Subcutaneous Injection: 5 x 2 μg
- 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose: OLP-1002 (Test): Part B, Multiple Ascending Dose: Subcutaneous Injection: 5 x 5 μg
- 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose: OLP-1002 (Test): Part B, Multiple Ascending Dose: Subcutaneous Injection: 5 x 10 μg
- 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose: OLP-1002 (Test): Part B, Multiple Ascending Dose: Subcutaneous Injection: 5 x 20 μg
- 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose: OLP-1002 (Test): Part B, Multiple Ascending Dose: Subcutaneous Injection: 5 x 40 μg
- 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose: OLP-1002 (Test): Part B, Multiple Ascending Dose: Subcutaneous Injection: 5 x 80 μg
Period: Overall Study
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Started | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose | Total
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 116
Age, Customized [Mean (Standard Deviation); unit: years] | 36.2 (12.25) | 35.7 (11.55) | 36.3 (10.44) | 37.0 (11.27) | 37.0 (14.25) | 44.0 (12.17) | 33.8 (11.97) | 34.0 (2.65) | 52.3 (6.35) | 43.7 (15.25) | 40.8 (11.27) | 43.5 (12.71) | 39.7 (10.75) | 35.7 (13.60) | 34.8 (13.70) | 41.0 (8.72) | 42.5 (11.31) | 37.3 (15.37) | 33.3 (13.92) | 38.4 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 2 | 2 | 2 | 1 | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 40
  Male | 11 | 2 | 4 | 3 | 4 | 3 | 5 | 1 | 1 | 4 | 4 | 5 | 8 | 3 | 4 | 3 | 4 | 2 | 5 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 5 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 115
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 7
  White | 14 | 3 | 5 | 3 | 5 | 3 | 5 | 2 | 3 | 5 | 5 | 6 | 11 | 4 | 5 | 4 | 5 | 6 | 6 | 100
  More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 175.2 (9.00) | 183.3 (12.06) | 177.3 (6.89) | 177.3 (6.51) | 173.8 (8.89) | 170.0 (6.00) | 174.2 (7.99) | 166.7 (3.79) | 173.0 (12.17) | 172.7 (9.31) | 176.0 (15.31) | 170.0 (5.44) | 177.1 (10.59) | 174.0 (12.81) | 175.3 (9.71) | 167.7 (6.65) | 173.2 (6.71) | 167.7 (12.53) | 176.8 (4.31) | 174.0 (9.33)
Body Weight [Mean (Standard Deviation); unit: kg] | 75.74 (11.677) | 77.47 (20.400) | 77.32 (9.601) | 75.33 (18.230) | 70.78 (8.725) | 73.80 (0.624) | 73.17 (6.910) | 66.00 (4.513) | 72.53 (11.441) | 72.72 (9.353) | 76.20 (15.517) | 72.23 (9.673) | 77.61 (8.632) | 73.03 (14.719) | 73.03 (14.844) | 64.08 (9.853) | 70.88 (9.658) | 67.02 (13.707) | 75.65 (9.408) | 73.37 (11.061)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.54 (2.410) | 22.73 (3.585) | 24.60 (2.649) | 23.73 (4.136) | 23.45 (2.421) | 25.63 (2.003) | 24.10 (1.439) | 23.73 (0.551) | 24.17 (2.335) | 24.43 (2.942) | 24.37 (1.279) | 24.95 (2.513) | 24.73 (1.512) | 23.95 (1.925) | 23.53 (2.642) | 22.70 (2.321) | 23.57 (1.941) | 23.70 (2.700) | 24.18 (2.780) | 24.13 (2.240)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Stratified by Overall and Severity
Description: Participants were observed for any signs or symptoms of adverse events and asked about their condition by open questioning, such as "How have you been feeling since you were last asked?", at least once each day while resident at the study site and at each study visit.
Time Frame: Part A: From screening through study completion, up to 32 days. Part B: From screening through study completion, up to 60 days.
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Treatment-emergent adverse events (Overall) | 7 | 3 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 5 | 3 | 7 | 3 | 4 | 5 | 4 | 6 | 5
  Mild | 6 | 3 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 5 | 3 | 7 | 3 | 4 | 4 | 3 | 6 | 5
  Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced Clinically Important Changes in Supine Diastolic and Systolic Blood Pressure
Description: Number of participants who experienced clinically important changes from baseline (the last value recorded prior to first dose) to scheduled timepoints in supine diastolic and systolic blood pressure.
  Participants were supine for at least 5 minutes before blood pressure measurements. Blood pressure was measured in triplicate and the time of measurement are below:
  Single ascending dose: Predose, 1, 2, 4, 8, 24 (± 1 hours), and 48 hours posdose Multiple ascending dose: Day 1 (Predose, 1, 2, 4, and 8 hours postdose), Day 2, Day 4 (postdose), Day 5, Day 7 (postdose), Day 9, Day 10 (postdose), Day 12, Day 13 (predose, 1, 2, 4, and 8 hours postdose), and Day 15
  No treatment or dose related trends and no clinically significant changes were observed in mean or individual participant supine blood pressure.
  Supine diastolic blood pressure reference range: 90 to 140 mmHg. Supine systolic blood pressure reference range: 50 to 90 mmHg.
Time Frame: as for outcome 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Diastolic blood pressure (mmHg) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic blood pressure (mmHg) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced Clinically Important Changes in Supine Pulse Rate
Description: Number of participants who experienced clinically important changes from baseline (the last value recorded prior to first dose) to scheduled timepoints in supine pulse rate.
  Participants were supine for at least 5 minutes before pulse rate measurements. Pulse rate was measured in triplicate and the time of measurement are below:
  Single ascending dose: Predose, 1, 2, 4, 8, 24 (± 1 hours), and 48 hours posdose Multiple ascending dose: Day 1 (Predose, 1, 2, 4, and 8 hours postdose), Day 2, Day 4 (postdose), Day 5, Day 7 (postdose), Day 9, Day 10 (postdose), Day 12, Day 13 (predose, 1, 2, 4, and 8 hours postdose), and Day 15
  No treatment or dose related trends and no clinically significant changes were observed in mean or individual participant supine pulse rate.
  Reference range: 40 to 100 beats per minute.
Time Frame: as for outcome 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced Clinically Important Changes in Respiratory Rate
Description: Number of participants who experienced clinically important changes from baseline (the last value recorded prior to first dose) to scheduled timepoints in respiratory rate.
  Participants were supine for at least 5 minutes before respiratory rate measurements. Respiratory rate was measured in triplicate and the time of measurement are below:
  Single ascending dose: Predose, 1, 2, 4, 8, 24 (± 1 hours), and 48 hours posdose Multiple ascending dose: Day 1 (Predose, 1, 2, 4, and 8 hours postdose), Day 2, Day 4 (postdose), Day 5, Day 7 (postdose), Day 9, Day 10 (postdose), Day 12, Day 13 (predose, 1, 2, 4, and 8 hours postdose), and Day 15
  No treatment or dose related trends and no clinically significant changes were observed in mean or individual participant respiratory rate.
  Reference range: 10 to 24 breaths per minute.
Time Frame: as for outcome 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: 12-lead Electrocardiogram Parameters
Description: Resting 12-lead electrocardiogram parameters were recorded after the participant had been supine and at rest for at least 5 minutes.
  Baseline: the last value recorded prior to first dose; QTcB: QT interval corrected for heart rate using Bazett's formula; QTcF: QT interval corrected for heart rate using Fridericia's method.
Time Frame: as for outcome 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Maximum postdose QTcB greater than 450 milliseconds | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Maximum increase from baseline in QTcB greater than 30 milliseconds | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 2
  Maximum postdose QTcF greater than 450 milliseconds | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Maximum increase from baseline in QTcF greater than 30 milliseconds | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0

6. Primary Outcome: Number of Participants With Findings of Clinical Importance in Clinical Chemistry, Hematology, and Urinalysis Test Results
Description: Number of participants with findings of clinical importance in clinical chemistry, hematology, and urinalysis test results.
  Clinical laboratory evaluations included:
  Clinical chemistry: Alanine aminotransferase; Albumin; Alkaline phosphatase; Aspartate aminotransferase; Calcium; Chloride; Cholesterol; Creatinine; Direct bilirubin; Gamma-glutamyl transferase; Glucose; Inorganic phosphate; Potassium; Sodium; Total bilirubin; Total protein; Urea Hematology: Hematocrit; Hemoglobin; Mean cell hemoglobin; Mean cell hemoglobin concentration; Mean cell volume; Platelet count; Red blood cell count; White blood cell count; White blood cell differential (Basophils; Eosinophils; Lymphocytes; Monocytes; Neutrophils) Urinalysis: Blood; Glucose; Ketones; pH; Protein; Specific gravity; Urobilinogen; Microscopic examination
Time Frame: as for outcome 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Full and Symptom-Directed Physical Examination Results
Description: A full physical examination and symptom-directed physical examinations were performed at specified timepoints.
Time Frame: as for outcome 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Medical device site rash (clinically significant, not related to study drug) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sunburn (clinically significant, not related to study drug) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Papule (clinically significant, not related to study drug) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Tongue ulceration (clinically significant, not related to study drug) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Gingival swelling (clinically significant, not related to study drug) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Injection Site Assessment Results
Description: Evaluation of the dosing site for the following:
  Pain: Grade 0 to 4 Redness (assessed by estimating the size of the red patch at the injection site across its widest point): Grade 0: 0-24 mm; Grade 1: 25-50 mm; Grade 2: 51-100 mm; Grade 3: More than 100 mm; Grade 4: Requires medical intervention greater than analgesia Swelling (assessed by estimating the size of the raised area around the injection site across its widest point): Grade 0: 0-24 mm; Grade 1: 25-50 mm and does not interfere with activity; Grade 2: 51-100 mm or interferes with activity; Grade 3: More than 100 mm and prevents daily activity; Grade 4: Requires medical intervention greater than analgesia Tenderness: Grade 0 to 4
  Bruising and ulceration were evaluated as present or absent.
Time Frame: as for outcome 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 17 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Pain : Grade 1 (does not interfere with activity) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Pain : Grade 2 (interferes with activity or repeated use of non-narcotic pain reliever) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tenderness : Grade 1 (mild pain to touch) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Tenderness : Grade 2 (moderate pain to touch) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness : Grade 1 (25-50 mm) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Redness : Grade 2 (51-100 mm) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling : Grade 1 (25-50 mm) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Swelling : Grade 2 (51-100 mm or interferes with activity) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising : Present | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 1

9. Primary Outcome: Number of Participants With Exposure to OLP-1002 That Exceeded Pre-define Exposure Limits From Non-clinical Studies
Description: Participants were assessed to demonstrate that exposure to OLP-1002 did not exceed pre-defined exposure limits from non-clinical studies. Participants with temporary detected plasma concentrations between the low limit of detection [0.2 ng/mL] and lower limit of quantification [1 ng/mL] are presented in the results.
Time Frame: Part A: Day 1 postdose. Part B: Day 1 postdose and Day 13 postdose.
Population: Safety Population.
  Plasma concentrations of OLP-1002 were not analyzed for the groups receiving single doses of 30 ng, 120 ng, 400 ng, 1.2 µg, and 3 µg OLP-1002 and were assumed also to be below the lower limit of quantification/limit of detection. Day 13 assessments were not applicable for Part A of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Day 1 Postdose: number analyzed (Participants) | 3 | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Day 1 Postdose | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0 | 3 | 6
  Day 13 Postdose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6
  Day 13 Postdose |  |  |  |  |  | 0 | 0 | 0 | 0 | 3 | 5

ADVERSE EVENTS:
Time Frame: Part A: From Screening until Poststudy (Day 28 ±2 days); Part B: From Screening until Poststudy (Day 57 ±2 days)
Description: The condition of each participant was monitored from the time of signing informed consent form to final discharge from the study. Participants were observed for any signs or symptoms and asked about their condition by open questioning, such as "How have you been feeling since you were last asked?", at least once each day while resident at the study site and at each study visit. Participants were also encouraged to spontaneously report adverse events occurring at any other time during the study.
Arm/Group | Placebo Part A, Single Ascending Dose | 30 ng OLP-1002: Part A, Single Ascending Dose | 120 ng OLP-1002: Part A, Single Ascending Dose | 400 ng OLP-1002: Part A, Single Ascending Dose | 1.2 µg OLP-1002: Part A, Single Ascending Dose | 3 µg OLP-1002: Part A, Single Ascending Dose | 6 µg OLP-1002: Part A, Single Ascending Dose | 12 µg OLP-1002: Part A, Single Ascending Dose | 20 µg OLP-1002: Part A, Single Ascending Dose | 40 µg OLP-1002: Part A, Single Ascending Dose | 80 µg OLP-1002: Part A, Single Ascending Dose | 160 µg OLP-1002: Part A, Single Ascending Dose | 5 x Placebo Part B, Multiple Ascending Dose | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/3 | 0/6 | 0/3 | 0/6 | 0/3 | 0/6 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/3 | 0/6 | 0/3 | 0/6 | 0/3 | 0/6 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 7/17 | 3/3 | 2/6 | 0/3 | 0/6 | 1/3 | 2/6 | 0/3 | 0/3 | 3/6 | 5/6 | 3/6 | 7/12 | 3/6 | 4/6 | 5/6 | 4/6 | 6/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Part A, Single Ascending Dose (N=17) | 30 ng OLP-1002: Part A, Single Ascending Dose (N=3) | 120 ng OLP-1002: Part A, Single Ascending Dose (N=6) | 400 ng OLP-1002: Part A, Single Ascending Dose (N=3) | 1.2 µg OLP-1002: Part A, Single Ascending Dose (N=6) | 3 µg OLP-1002: Part A, Single Ascending Dose (N=3) | 6 µg OLP-1002: Part A, Single Ascending Dose (N=6) | 12 µg OLP-1002: Part A, Single Ascending Dose (N=3) | 20 µg OLP-1002: Part A, Single Ascending Dose (N=3) | 40 µg OLP-1002: Part A, Single Ascending Dose (N=6) | 80 µg OLP-1002: Part A, Single Ascending Dose (N=6) | 160 µg OLP-1002: Part A, Single Ascending Dose (N=6) | 5 x Placebo Part B, Multiple Ascending Dose (N=12) | 5 x 2 μg OLP-1002: Part B, Multiple Ascending Dose (N=6) | 5 x 5 μg OLP-1002: Part B, Multiple Ascending Dose (N=6) | 5 x 10 μg OLP-1002: Part B, Multiple Ascending Dose (N=6) | 5 x 20 μg OLP-1002: Part B, Multiple Ascending Dose (N=6) | 5 x 40 μg OLP-1002: Part B, Multiple Ascending Dose (N=6) | 5 x 80 μg OLP-1002: Part B, Multiple Ascending Dose (N=6)
Headache (Nervous system disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site rash (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — General disorders and administration site conditions
Infusion site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Medical device site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Medical device site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Medical device site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 — General disorders and administration site conditions
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — General disorders and administration site conditions
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — General disorders and administration site conditions
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — General disorders and administration site conditions
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall not use the name, trademark or the name of any representative of the other, or the existence of their agreement with the sponsor for any promotional or advertising purposes, or any other publication, without the prior written consent of the sponsor, or state or imply that the sponsor endorses or approves any service, material, product or compound of the sponsor without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT03760913/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03760913/SAP_001.pdf